CLINICAL TRIAL: NCT05472142
Title: Clinical Trial Protocol: Using Practice Facilitation and Operationalizing Referral Information Technology (UP FOR IT) to Increase DSMES Utilization
Brief Title: Using Practice Facilitation and Operationalizing Referral Information Technology to Increase DSMES Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Lacy (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Mary Lacy, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 75928; R34DK132548 (NIH)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Diabetes
Keywords: diabetes self-management education and support (DSMES); implementation science; practice facilitation; health information technology; evidence-based practice; rural clinics
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Cluster (Active Comparator): Clinics in the control group will only be provided with health information technology; they will not participate in the 12-month intervention which incorporates health information technology and practice facilitation.
  Interventions: Other: UP FOR IT - health information technology
- Intervention Cluster (Experimental): Clinics in the intervention group will participate in the 12-month intervention which incorporates health information technology and practice facilitation.
  Interventions: Other: UP FOR IT - practice facilitation; Other: UP FOR IT - health information technology

INTERVENTIONS:
Other: UP FOR IT - practice facilitation — Using Practice Facilitation and Operationalizing Referral Information Technology (UP FOR IT) involves incorporation of health information technology and practice facilitation. The practice facilitation collaborative trains and supports clinical teams to use the Model for Improvement to make "breakthrough" improvements in diabetes care and DSMES utilization by recognizing barriers and changing clinical systems and care practices.
  Arms: Intervention Cluster
Other: UP FOR IT - health information technology — Using Practice Facilitation and Operationalizing Referral Information Technology (UP FOR IT) involves incorporation of health information technology and practice facilitation. The health information technology component provides the scaffolding for quality improvement efforts by automating patient identification and enabling bi-directional referral communication between providers and diabetes self-management education and services (DSMES) programs.

SUMMARY:
This is a pilot and feasibility study of a pragmatic cluster randomized trial that utilizes health information technology and practice facilitation to address referral barriers and increase clinician awareness and motivation to refer patients with diabetes to diabetes self-management education and services (DSMES).

DETAILED DESCRIPTION:
Diabetes self-management education and support (DSMES) is an evidence-based educational program that helps people with diabetes better control their blood sugar (improved hemoglobin A1c) and reduce diabetes-related complications and healthcare costs. DSMES is strikingly underutilized with fewer than 10% of eligible patients receiving this helpful service due to patient-, clinician-, and health system-level barriers that include low clinician awareness and lack of integrated referral processes between clinics and community-based DSMES programs.

In this study, we will conduct a pilot and feasibility study of a pragmatic cluster randomized trial that utilizes health information technology and practice facilitation to address referral barriers and increase clinician awareness and motivation to refer patients with diabetes to DSMES. We have partnered with the Kentucky Department of Public Health (KDPH, statewide DSMES provider), the Kentucky Regional Extension Center (KY-REC, practice facilitation partner), and the Kentucky Health Information Exchange (health information technology (HIT) partner). We will recruit two healthcare systems in rural Kentucky to participate in the study. Within each healthcare organization, we will randomize control and intervention clusters at the clinic level. Clinics in the intervention group will participate in the 12-month intervention which incorporates health information technology and practice facilitation. The health information technology component provides the scaffolding for quality improvement efforts by automating patient identification and enabling bi-directional referral communication between providers and DSMES programs. Health information technology support will be available at all clinic sites within participating health care organizations, including the control clinics. The practice facilitation collaborative trains and supports clinical teams to use the Model for Improvement to make "breakthrough" improvements in diabetes care and DSMES utilization by recognizing barriers and changing clinical systems and care practices.

ELIGIBILITY:
Inclusion Criteria:

- Clinics are being recruited to participate in the intervention. All clinic staff at participating clinics are eligible for inclusion in the study.

Exclusion Criteria:

- There are no exclusion criteria beyond employment at a participating clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lacy, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentukcy, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We partnered with two healthcare systems in rural Kentucky to test a pragmatic cluster-randomized trial. Within each healthcare system, we identified three primary care clinics that had a sufficient volume (N>50) of patients age 18-75 with diabetes. We randomized two of the clinics within each healthcare system to the intervention arm (total intervention clinics = 4) and one to the control arm (total control clinics =2).
Pre-assignment Details: Study participants included clinic staff (n=22 total, consented) and patients (n=1,803, not consented). Clinic staff received the intervention and patients of clinics could be indirectly impacted by intervention. Clinic staff aggregated patient data up to the clinic-level prior to sharing with the study team. Patients were not consented as there was no interaction from members of the research team with patients and there was no use of identifiable private information for research purposes.
Units Other Than Participants: Clinics
Groups:
- Arm: Control Clinic: Control clinic level
- Arm: Intervention Clinic: Intervention Clinic Level
Period: Total Participants
Arm/Group | Arm: Control Clinic | Arm: Intervention Clinic
Started | 726; 2 Clinics | 1099; 4 Clinics
Completed | 414; 2 Clinics | 1099; 4 Clinics
Not Completed | 312; 0 Clinics | 0; 0 Clinics
Not completed — Lost to Follow-up | 312 | 0
Period: Clinic Patients
Arm/Group | Arm: Control Clinic | Arm: Intervention Clinic
Started | 720; 2 Clinics | 1083; 4 Clinics
Completed | 408; 2 Clinics | 1083; 4 Clinics
Not Completed | 312; 0 Clinics | 0; 0 Clinics
Not completed — Lost to Follow-up | 312 | 0
Period: Clinic Staff
Arm/Group | Arm: Control Clinic | Arm: Intervention Clinic
Started | 6; 2 Clinics | 16; 4 Clinics
Completed | 6; 2 Clinics | 16; 4 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Arm: Control Cluster: Active Comparator - number of participants
- Arm: Intervention Cluster: Experimental - number of participants
- Total: Total of all reporting groups
Arm/Group | Arm: Control Cluster | Arm: Intervention Cluster | Total
Number analyzed (Participants) | 726 | 1099 | 1825
Age, Customized [Count of Participants; unit: Participants] — Population: The Row populations differs from the Overall population because there are two distinct populations that, together, make up the Overall population - clinic staff and patients.
  Participants
    Clinic staff: number analyzed (Participants) | 6 | 16 | 22
    Clinic staff: <18 years old | 0 | 0 | 0
    Clinic staff: 18-75 years old | 6 | 16 | 22
    Clinic staff: >75 years old | 0 | 0 | 0
    Patients: number analyzed (Participants) | 720 | 1083 | 1803
    Patients: <18 years old | 0 | 0 | 0
    Patients: 18-75 years old | 720 | 1083 | 1803
    Patients: >75 years old | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Row populations differs from the Overall population because there are two distinct populations that, together, make up the Overall population - clinic staff and patients.
  Participants
    Clinic Staff: number analyzed (Participants) | 6 | 16 | 22
    Clinic Staff: Female | 6 | 15 | 21
    Clinic Staff: Male | 0 | 1 | 1
    Patients: number analyzed (Participants) | 720 | 1083 | 1803
    Patients: Female | 700 | 1000 | 1700
    Patients: Male | 20 | 83 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Row populations differs from the Overall population because there are two distinct populations that, together, make up the Overall population - clinic staff and patients.
  Participants
    Clinic Staff: number analyzed (Participants) | 6 | 16 | 22
    Clinic Staff: Hispanic or Latino | 0 | 0 | 0
    Clinic Staff: Not Hispanic or Latino | 6 | 16 | 22
    Clinic Staff: Unknown or Not Reported | 0 | 0 | 0
    Patients: number analyzed (Participants) | 720 | 1083 | 1803
    Patients: Hispanic or Latino | 0 | 6 | 6
    Patients: Not Hispanic or Latino | 720 | 1065 | 1785
    Patients: Unknown or Not Reported | 0 | 12 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Row populations differs from the Overall population because there are two distinct populations that, together, make up the Overall population - clinic staff and patients.
  Participants
    Clinic Staff: number analyzed (Participants) | 6 | 16 | 22
    Clinic Staff: American Indian or Alaska Native | 0 | 0 | 0
    Clinic Staff: Asian | 0 | 0 | 0
    Clinic Staff: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Clinic Staff: Black or African American | 0 | 0 | 0
    Clinic Staff: White | 6 | 16 | 22
    Clinic Staff: More than one race | 0 | 0 | 0
    Clinic Staff: Unknown or Not Reported | 0 | 0 | 0
    Patients: number analyzed (Participants) | 720 | 1083 | 1803
    Patients: American Indian or Alaska Native | 0 | 0 | 0
    Patients: Asian | 1 | 1 | 2
    Patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patients: Black or African American | 1 | 6 | 7
    Patients: White | 702 | 1064 | 1766
    Patients: More than one race | 0 | 0 | 0
    Patients: Unknown or Not Reported | 16 | 12 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 726 | 1099 | 1825
Diabetes Self-Management Education & Support referral during 12-month baseline period [Count of Participants; unit: Participants] — Population: The analysis population differs from the Overall population because the study has two distinct populations that, together, make up the Overall population - clinic staff and patients. This study-specific baseline measure was only captured on one of the two populations - patients.
  Participants
    number analyzed (Participants) | 720 | 1083 | 1803
    Referred to DSMES | 0 | 0 | 0
    Not referred to DSMES | 720 | 1083 | 1803
Percent of patient population with A1c >9% at baseline [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: The analysis population differs from the Overall population because the study has two distinct populations that, together, make up the Overall population - clinic staff and patients. This study-specific baseline measure was only captured on one of the two populations - patients.
  Participants
    number analyzed (Participants) | 720 | 1083 | 1803
    A1c greater than 9% | 149 | 206 | 355
    A1c less than or equal to 9% | 571 | 877 | 1448

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Self-Management Education and Support (DSMES) Referrals
Description: DSMES referrals will be measured as the referral rate at baseline, the end of the active intervention and the end of the follow-up period. The outcome will be assessed through clinic electronic health record data.
Time Frame: Baseline, End of active intervention (month 9), End of follow-up (month 15)
Population: Measure Analysis Population Description: The analysis population differs from the Overall population because the study has two distinct populations that, together, make up the Overall population - clinic staff and patients. This study-specific baseline measure was only captured on one of the two populations - patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm: Control Cluster | Arm: Intervention Cluster
Number analyzed (Participants) | 720 | 1083
Participants
  Baseline | 0 | 0
  End of active intervention | 4 | 343
  End of follow-up | 4 | 433

2. Secondary Outcome: Diabetes Self-Management Education and Support (DSMES) Attendance
Description: DSMES attendance will be measured as DSMES attendance rate at baseline, the end of the active intervention and the end of follow-up period. The outcome will be assessed through aggregated, de-identified data that is routinely collected by DSMES providers.
Time Frame: Baseline, End of active intervention (month 9), End of follow-up (month 15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm: Control Cluster | Arm: Intervention Cluster
Number analyzed (Participants) | 720 | 1083
Participants
  Baseline | 0 | 0
  End of active intervention | 0 | 22
  End of follow-up | 0 | 61

3. Secondary Outcome: Percent of Patients With A1c >9%
Description: Percent of patients with A1c >9% at baseline, the end of the active intervention and the end of follow-up period. The outcome will be assessed through clinic-level aggregate data extracted from electronic health record data.
Time Frame: Baseline, End of active intervention (month 9), End of follow-up (month 15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm: Control Cluster | Arm: Intervention Cluster
Number analyzed (Participants) | 720 | 1083
Participants
  Baseline | 149 | 206
  End of active intervention: number analyzed (Participants) | 408 | 1083
  End of active intervention | 93 | 194
  End of follow-up: number analyzed (Participants) | 408 | 1083
  End of follow-up | 93 | 173

ADVERSE EVENTS:
Description: Adverse events were not monitored/assessed for clinic staff or patients
Arm/Group | Arm: Control Cluster | Arm: Intervention Cluster
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT05472142/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT05472142/ICF_000.pdf